CLINICAL TRIAL: NCT04949984
Title: Bright Light Therapy in Older Adults With Moderate to Very Severe Dementia: Effects on Cognition, Mood, Behavior, and Physiological Parameters
Brief Title: Bright Light Therapy in Older Adults With Moderate to Very Severe Dementia
Acronym: BLT-Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, José Carlos Millán Calenti, Full Professor, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/408; ED431C 2017/49 (Other Grant/Funding Number: Xunta de Galicia); ED431F 2017/09 (Other Grant/Funding Number: Xunta de Galicia); IN607C 2016/08 (Other Grant/Funding Number: Xunta de Galicia); IN607C 2017/02 (Other Grant/Funding Number: Xunta de Galicia); RYC-2015-18394 (Other Grant/Funding Number: Spanish Ministry of Economy and Competitiveness)
Record Dates: First submitted 2021-06-18; First posted 2021-07-02 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Dementia; Mood; Behavior
Keywords: bright light therapy; oxygen saturation; heart rate
MeSH Terms: conditions — Dementia; Behavior | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright light therapy (Experimental): The devices used for the intervention were bright white light lamps providing an intensity of 10,000 lux. Four users participated in each session, placing two users per lamp, seated in a comfortable chair with armrests 70 cm from the lamp. The sessions were 30 minutes/day in the time slot between 10:30 and 12:00 in the morning, 5 days a week (Monday to Friday) for 4 weeks (total 20 sessions). Two groups of participants per day were established, the first shift being from 10:30 to 11:00, and the second from 11:15 to 11:45 a.m., which means the stimulation of 8 people per day (month). During the sessions, while exposed to light, participants were watching documentaries on neutral topics (nature, Spanish and Galician culture, etc.).
  Interventions: Device: Bright light therapy
- Control group (No Intervention): Participants were evaluated before and after the experimental group finishes the intervention program (pre- vs. postintervention) to facilitate an examination of the changes in the outcome measures.

INTERVENTIONS:
Device: Bright light therapy — BLT consisted of 30-minute morning sessions with an intensity of 10,000 lux, five days a week (Monday to Friday), for 4 weeks.
  Other Names: BLT
  Arms: Bright light therapy

SUMMARY:
INTRODUCTION: Bright light therapy (BLT) has demonstrated positive effects on sleep, mood, and behavioral problems in older adults with dementia. However, there is little research in people with advanced stages of dementia.

OBJECTIVES: Main objectives are to study the immediate effects, short and long-term effects of BLT in a sample of institutionalized older adults with moderate to very severe dementia. Later, to compare the potential effectiveness of bright light therapy sessions with other non-pharmacological interventions in people with dementia.

METHODS AND ANALYSIS: The study was a 2 x 2 randomized controlled trial using a two-group design (BLT vs. control) and two repeated measures (pre- vs. postintervention). In addition, the BLT group participants were assessed immediately before, after, and during each session. The BLT protocol consisted of 30-minute morning sessions of 10,000 lux, Monday through Friday, for 4 weeks.

For the statistical analysis, two-way analysis of variance (ANOVA) are used to determine the existence of differences at two points in time (pre- vs. post-). The Wilcoxon signed-rank test or the Paired t test are used to measure changes from before to after the intervention sessions.

DETAILED DESCRIPTION:
INTRODUCTION: Dementia is one of the main causes of disability and dependence among older adults worldwide, constituting a public health priority due to its significant human and financial costs to society. Pharmacological and non-pharmacological interventions have been proposed for the management of its clinical manifestations. The nonpharmacological interventions, which include bright light therapy (BLT), are recommended by numerous guidelines as initial treatment strategies due to the absence of adverse events. BLT consists of the controlled application of certain levels of light that can be administered in several ways. There is some evidence that effective doses of light would stimulate circadian cycles, thus affecting sleep efficiency, depression, or behavioral problems in older adults with dementia, but there is little research on persons in advanced stages of dementia.

The lack of consensus on the protocol for BLT application, as well as the existence of little research on individuals in advanced stages of dementia, calls for further research to explore in-depth the immediate, short- and long-term effects of BLT in this population.

OBJECTIVES: Main objectives were: (1) to study the short- and long-term effects of bright light therapy on mood, behavior, sleep, and cognition in a sample of institutionalized older adults with moderate to very severe dementia; (2) to explore the immediate effects of bright light therapy sessions on behavior, mood and physiological parameters in a sample of institutionalized older adults with moderate to very severe dementia; and (3) to compare the effectiveness of bright light therapy sessions with other non-pharmacological interventions in people with dementia.

METHODS: This longitudinal, comparative and prospective study, is a 2 x 2 randomized controlled trial using a two-group design (BLT vs. control) and two repeated measures (pre- vs. postintervention). In addition, the BLT group participants were assessed immediately before, after, and during each session. Participants were recruited among residents of the Gerontological Complex La Milagrosa (A Coruña, Spain). The BLT protocol consisted of 30-minute morning sessions in the time slot between 10:30 and 12:00, 5 days a week (Monday to Friday), for 4 weeks (total 20 sessions). The devices used for the intervention were bright white light lamps providing an intensity of 10,000 lux. Four users participated in each session, placing two users per lamp, seated 70 cm from the lamp. All data analysis will be performed with the statistical programs SPSS- Statistical Package for the Social Sciences (version 25.0), RStudio software package (Version 1.3.1093), and JAMOVI (The jamovi project, 2020, Version 1.2).

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* diagnosis of dementia
* a score ≥ 4 points on the Global Deterioration Scale (GDS; Reisberg et al., 1982), ranging from moderate to very severe cognitive decline.

Exclusion Criteria:

* high ocular sensitivity to light (photosensitivity)
* preexisting ocular abnormalities
* having any severe ocular disorder that did not allow them to open their eyes or that implied a very low visual acuity.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Age | 4 weeks
  Age (years), including the birth date.
Gender | 4 weeks
  Male or female.
Educational level | 4 weeks
  Number of years of education (≤ 8, 9-17 or >17)
Cognitive status- Screening | 4 weeks
  Mini-Mental State Examination (MMSE). Cognitive evaluation: a brief screening test for cognitive impairment. MMSE is a 30-point test, in which lower scores mean worse cognitive status. The cut-off point for determining the presence of cognitive impairment is normally set at 24 points.
Severe cognitive status- Screening | 4 weeks
  Severe Mini-Mental State Examination (SMMSE). Cognitive evaluation: brief assessment of severe cognitive impairment in advanced stages of dementia. This test was applied only to individuals who obtained a score of 10 points or less in the MMSE. SMMSE, totals 30 points, lower scores mean worse cognitive status.
Cognitive status- Level | 4 weeks
  Cambridge Cognitive Examination (CAMCOG). Cognitive evaluation: more comprehensive cognitive assessment of participants with moderate cognitive impairment (GDS = 4). This scale includes the evaluation of the following domains: orientation, language, memory, attention and calculation, praxis, abstraction, perception and executive function. CAMCOG is a 107- point scale and scores of less than 80 have been suggested as cut-off for dementia.
Cognitive domains | 4 weeks
  Severe Cognitive Impairment Profile (SCIP). Cognitive evaluation: a more comprehensive cognitive assessment of participants with moderate-severe to very severe cognitive impairment (GDS = 5, 6 and 7). This scale allows obtaining a performance profile in each of the cognitive domains evaluated (comportment, attention, language, memory, motor, conceptualization, arithmetic, and visuospatial) and calculating a total score indicative of the degree of cognitive impairment: moderately severe, severe, very severe and profound. Higher scores mean higher cognitive impairment.
Depression in Dementia | 4 weeks
  The Cornell Scale for Depression in Dementia (CSDD). Mood evaluation: assessment of signs and symptoms of major depression in patients with dementia focusing on the week preceding the interview. The Cornell Scale utilizes two semi-structured comprehensive interviews that elicits information from the patient and the informant. In those cases in which the patient is not able to respond due to the level of cognitive impairment, information is obtained only from the interview with the informant. Total score ranges from 0 to 38; above 10 indicate a probable major depression and above 18 indicates a definite major depression.
Mood and behaviour | 4 weeks
  Neuropsychiatric Inventory Questionnaire (NPI-Q). Mood and behavior evaluation: a brief retrospective (1 month) caregiver self-administered questionnaire to assess caregiver distress and severity of 12 neuropsychiatric symptoms: delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviors, nighttime behavioral disturbances, and appetite/eating disturbances. For each of the symptoms the informant rates both its severity on a 3-point scale and the associated caregiver distress on a 5-point scale. The NPI-Q provides symptom severity and distress ratings for each symptom reported, and scores for total severity (0 to 36 points) and total distress (0 to 60 points) reflecting the sum of individual domain scores. Higher scores indicate higher severity and caregiver distress.
Agitation | 4 weeks
  Cohen-Mansfield Agitation Inventory (CMAI). Mood and behavior evaluation: a caregiver rating questionnaire for the assessment of the frequency of manifestations of agitated behaviors. Ratings refer to the two weeks prior to its administration. The CMAI consists of 29 agitated behaviors, each rated on a 7-point frequency scale (ranging from 1-Never to 7-Several times an hour), with higher scores indicating more agitation.
Anxiety | 4 weeks
  Rating for Anxiety in Dementia (RAID). Mood and behavior evaluation: a clinical rating scale to evaluate severity of anxiety including somatic symptoms and specific fears. Scoring should be based on the two weeks prior to the caregiver interview. The total score ranges from 0 to 40, with higher scores implying greater severity of anxiety disorder.
Sleep-disturbed behaviours | 4 weeks
  Sleep Disorders Inventory (SDI). Sleep evaluation: this inventory is an expanded version of one item of the Neuropsychiatric Inventory (NPI). It records the frequency (ranging from 0 to 4), the severity (from 0 to 3), and the caregiver distress (from 0 to 5) with respect to eight sleep-disturbed behaviors referred to the two weeks prior to its administration. Higher SDI scores mean greater frequency and severity of sleep disturbances.
Sleep-Actigraphy | 4 weeks
  Actiwatch AW4 - Actigraphy. Sleep evaluation: actigraphy is a non-invasive method of monitoring circadian rhythm. Actiwatchs are worn on the non-dominant wrist of the participants and record movements that are used to estimate sleep parameters with specialized algorithms in computer software programs. Both experimental and control group participants wore the actiwatch for 5 days before and 5 days after the intervention.
  Among the parameters obtained from actigraphy records, the following were chosen for analysis in the present study: sleep latency, sleep efficiency and total sleep
Disease severity in advanced stages of dementia. | 4 weeks
  Bedford Alzheimer Nursing Severity Scale (BANS-S). Functional evaluation: a nursing-staff administered questionnaire for the assessment of disease severity in advanced stages of dementia. The questionnaire comprises 7 items: dressing, sleep-wake cycle disturbances, speech, eating, ambulating, muscle rigidity and eye contact. BANS-S total score ranges from 7 to 28 and higher scores means higher dementia severity.
Mood and behaviour during, preceding and immediately after the sessions | 4 weeks
  Interact scale. Mood and behavior evaluation: the Interact Scale, and its shortened version, named Interact short, were used for the evaluation of immediate effects in the experimental group. Both allow the assessment of changes in mood and behavior, the Interact scale during the sessions, and the Interact short scale in the 10 minutes immediately preceding and in the 10 minutes immediately following the session. Each of the items is evaluated on a 5-option answer scale ranging from "not al all" to "Nearly all the time". Higher scores mean a higher frequency of occurrence of each type of mood and behavior evaluated.
Mean Heart rate | 4 weeks
  The baseline hemodynamic state is characterized by storing the mean of the three lowest values for thirty seconds of heart rate (HRrest; in BPM, beats per minute) with a finger pulse oximeter.
Percentage of Oxygen saturation | 4 weeks
  Blood oxygen saturation (%) of the participants in the experimental group is recorded at the beginning and end of each session using a mobile finger pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: José C. Millán-Calenti, Principal Investigator — Universidade da Coruña
Locations (1):
- Universidade da Coruña, A Coruña, Spain

REFERENCES:
- [Background] Abraha I, Rimland JM, Trotta FM, Dell'Aquila G, Cruz-Jentoft A, Petrovic M, Gudmundsson A, Soiza R, O'Mahony D, Guaita A, Cherubini A. Systematic review of systematic reviews of non-pharmacological interventions to treat behavioural disturbances in older patients with dementia. The SENATOR-OnTop series. BMJ Open. 2017 Mar 16;7(3):e012759. doi: 10.1136/bmjopen-2016-012759. PMID 28302633
- [Background] Dyer SM, Harrison SL, Laver K, Whitehead C, Crotty M. An overview of systematic reviews of pharmacological and non-pharmacological interventions for the treatment of behavioral and psychological symptoms of dementia. Int Psychogeriatr. 2018 Mar;30(3):295-309. doi: 10.1017/S1041610217002344. Epub 2017 Nov 16. PMID 29143695
- [Background] Forbes D, Blake CM, Thiessen EJ, Peacock S, Hawranik P. Light therapy for improving cognition, activities of daily living, sleep, challenging behaviour, and psychiatric disturbances in dementia. Cochrane Database Syst Rev. 2014 Feb 26;2014(2):CD003946. doi: 10.1002/14651858.CD003946.pub4. PMID 24574061
- [Background] Lyketsos CG, Steinberg M, Tschanz JT, Norton MC, Steffens DC, Breitner JC. Mental and behavioral disturbances in dementia: findings from the Cache County Study on Memory in Aging. Am J Psychiatry. 2000 May;157(5):708-14. doi: 10.1176/appi.ajp.157.5.708. PMID 10784462
- [Background] Sloane PD, Figueiro M, Cohen L. Light as Therapy for Sleep Disorders and Depression in Older Adults. Clin Geriatr. 2008 Mar 1;16(3):25-31. No abstract available. PMID 24285919
- [Background] Steinberg M, Shao H, Zandi P, Lyketsos CG, Welsh-Bohmer KA, Norton MC, Breitner JC, Steffens DC, Tschanz JT; Cache County Investigators. Point and 5-year period prevalence of neuropsychiatric symptoms in dementia: the Cache County Study. Int J Geriatr Psychiatry. 2008 Feb;23(2):170-7. doi: 10.1002/gps.1858. PMID 17607801
- [Background] van Maanen A, Meijer AM, van der Heijden KB, Oort FJ. The effects of light therapy on sleep problems: A systematic review and meta-analysis. Sleep Med Rev. 2016 Oct;29:52-62. doi: 10.1016/j.smrv.2015.08.009. Epub 2015 Sep 9. PMID 26606319
- [Derived] Cibeira N, Maseda A, Lorenzo-Lopez L, Gonzalez-Abraldes I, Lopez-Lopez R, Rodriguez-Villamil JL, Millan-Calenti JC. Bright Light Therapy in Older Adults with Moderate to Very Severe Dementia: Immediate Effects on Behavior, Mood, and Physiological Parameters. Healthcare (Basel). 2021 Aug 19;9(8):1065. doi: 10.3390/healthcare9081065. PMID 34442202

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT04949984/SAP_000.pdf